CLINICAL TRIAL: NCT04408638
Title: A Phase III, Open-Label, Multicenter, Randomized Study Evaluating the Efficacy and Safety of Glofitamab in Combination With Gemcitabine Plus Oxaliplatin Versus Rituximab in Combination With Gemcitabine and Oxaliplatin in Patients With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Phase III Study Evaluating Glofitamab in Combination With Gemcitabine + Oxaliplatin vs Rituximab in Combination With Gemcitabine + Oxaliplatin in Participants With Relapsed/Refractory Diffuse Large B-Cell Lymphoma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO41944; 2020-001021-31 (EudraCT Number)
Record Dates: First submitted 2020-05-26; First posted 2020-05-29 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — obinutuzumab; glofitamab; tocilizumab; Gemcitabine; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Glofit-GemOx (Experimental): Participants will receive up to 8 cycles of glofitamab (Glofit) in combination with gemcitabine and oxaliplatin (GemOx), followed by up to 4 cycles of glofitamab monotherapy. A single dose of obinutuzumab will be administered 7 days prior to the first dose of glofitamab. Treatment is administered in 21-day cycles.
  Interventions: Drug: Obinutuzumab; Drug: Glofitamab; Drug: Tocilizumab; Drug: Gemcitabine; Drug: Oxaliplatin
- R-GemOx (Experimental): Participants will receive rituxumab (R) in combination with gemcitabine and oxaliplatin (GemOx) for up to 8 cycles. Treatment is administered in 21-day cycles.
  Interventions: Drug: Rituxumab; Drug: Gemcitabine; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Obinutuzumab — Participants will receive a single dose of intravenous (IV) obinutuzumab pre-treatment 7 days prior to the first dose of glofitamab.
  Arms: Glofit-GemOx
Drug: Glofitamab — Participants will receive IV glofitamab for up to 12 cycles.
  Arms: Glofit-GemOx
Drug: Rituxumab — Participants will receive IV rituxumab on Day 1 of each cycle for up to 8 cycles.
  Arms: R-GemOx
Drug: Tocilizumab — Participants will receive IV tocilizumab as needed for treatment of cytokine-release syndrome (CRS).
  Arms: Glofit-GemOx
Drug: Gemcitabine — Participants will receive IV gemcitabine prior to oxaliplatin administration for up to 8 cycles.
Drug: Oxaliplatin — Participants will receive IV oxaliplatin after gemcitabine administration for up to 8 cycles.

SUMMARY:
This study will evaluate the efficacy and safety of glofitamab in combination with gemcitabine plus oxaliplatin (Glofit-GemOx) compared with rituximab in combination with gemcitabine plus oxaliplatin (R-GemOx) in patients with R/R DLBCL.

ELIGIBILITY:
Inclusion Criteria

* Histologically confirmed diffuse large B-cell lymphoma (DLBCL), not otherwise specified
* Relapsed/refractory (R/R) disease, defined as follows: Relapsed = disease that has recurred ≥6 months after completion of the last line of therapy; Refractory = disease that either progressed during the last line of therapy or progressed within 6 months (<6 months) of the last line of prior therapy
* At least one (≥1) line of prior systemic therapy
* Participants who have failed only one prior line of therapy must not be a candidate for high-dose chemotherapy followed by autologous stem cell transplant, as defined by the study protocol
* Confirmed availability of tumor tissue, unless unobtainable per investigator assessment. Freshly collected biopsy is preferred. Archival tissue is acceptable
* At least one bi-dimensionally measurable (≥1.5 cm) nodal lesion, or one bi-dimensionally measurable (≥1 cm) extranodal lesion, as measured on computed tomography (CT) scan
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0, 1, or 2
* Adequate hematologic function (unless attributable to the underlying disease, as established by extensive bone marrow involvement or associated with hypersplenism secondary to the involvement of the spleen by DLBCL per the investigator), as defined by the study protocol
* Negative SARS-CoV-2 antigen or PCR test within 7 days prior to enrollment
* Adequate renal function, defined as an estimated creatinine clearance ≥30 mL/min

Exclusion Criteria

* Patient has failed only one prior line of therapy and is a candidate for stem cell transplantation
* History of transformation of indolent disease to DLBCL
* High-grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements, and high-grade B-cell lymphoma not otherwise specified, as defined by 2016 WHO guidelines
* Primary mediastinal B-cell lymphoma
* History of severe allergic or anaphylactic reactions to humanized or murine monoclonal antibodies (or recombinant antibody-related fusion proteins) or known sensitivity or allergy to murine products
* Contraindication to obinutuzumab, rituximab, gemcitabine or oxaliplatin, or tocilizumab
* Prior treatment with glofitamab or other bispecific antibodies targeting both CD20 and CD3
* Peripheral neuropathy assessed to be Grade >1 according to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0 at enrollment
* Treatment with radiotherapy, chemotherapy, immunotherapy, immunosuppressive therapy, or any investigational agent for the purposes of treating cancer within 2 weeks prior to first study treatment
* Treatment with monoclonal antibodies for the purposes of treating cancer within 4 weeks prior to first study treatment
* Primary or secondary central nervous system (CNS) lymphoma at the time of recruitment or history of CNS lymphoma
* Current or history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment or any major episode of infection (as evaluated by the investigator) within 4 weeks prior to the first study treatment
* Positive SARS-CoV-2 infection within 30 days prior to the first study treatment, including asymptomatic SARS-CoV-2 infection
* Documented SARS-CoV-2 infection within 6 months of first study treatment
* Suspected or latent tuberculosis
* Positive for hepatitis B virus (HBV), hepatitis C virus (HCV), or human immunodeficiency virus (HIV)
* Known or suspected chronic active Epstein-Barr viral infection
* Known or suspected history of hemophagocytic lymphohistiocytosis (HLH)
* Known history of progressive multifocal leukoencephalopathy
* Adverse events from prior anti-cancer therapy not resolved to Grade 1 or better (with the exception of alopecia and anorexia)
* Administration of a live, attenuated vaccine within 4 weeks before first study treatment administration or anticipation that such a live, attenuated vaccine will be required during the study
* Prior solid organ transplantation
* Prior allogeneic stem cell transplant
* Active autoimmune disease requiring treatment
* Prior treatment with systemic immunosuppressive medications (including, but not limited to, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor agents), within 4 weeks prior to first dose of study treatment
* Corticosteroid therapy within 2 weeks prior to first dose of study treatment (exceptions defined by study protocol)
* Recent major surgery (within 4 weeks before the first study treatment) other than for diagnosis
* Clinically significant history of cirrhotic liver disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2021-02-23 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2028-03-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS), defined as the time from randomization to date of death from any cause | Up to 5 years

SECONDARY OUTCOMES:
Progression-free survival (PFS), defined as the time from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first, as determined by the Independent Review Committee (IRC) | Up to 5 years
PFS, defined as the time from randomization to the first occurrence of disease progression or death from any cause, whichever occurs first, as determined by the investigator | Up to 5 years
Complete response (CR) rate, defined as the proportion of patients whose best overall response is a CR on positron emission tomography/computed tomography (PET/CT) during the study, as determined by the IRC | Up to 5 years
CR rate, defined as the proportion of patients whose best overall response is a CR on positron emission tomography/computed tomography (PET/CT) during the study, as determined by the investigator | Up to 5 years
Objective response rate (ORR), defined as the proportion of patients whose best overall response is a partial response (PR) or a CR during the study, as determined by the IRC | Up to 5 years
ORR, defined as the proportion of patients whose best overall response is a partial response (PR) or a CR during the study, as determined by the investigator | Up to 5 years
Duration of objective response (DOR), defined as the time from the first occurrence of a documented objective response (CR or PR) to disease progression, or death from any cause, whichever occurs first | Up to 5 years
Duration of CR, defined as the time from the first occurrence of a documented CR to disease progression, or death from any cause, whichever occurs first | Up to 5 years
Time to deterioration in physical functioning and fatigue, as measured by the European Organisation for Research and Treatment of Cancer Quality of Life-Core 30 Questionnaire (EORTC QLQ-C30) | Up to 5 years
Time to deterioration in lymphoma symptoms, as measured by the Functional Assessment of Cancer Therapy-Lymphoma subscale (FACT-Lym LymS) | Up to 5 years
Percentage of Participants with Adverse Events | Up to 5 years
Tolerability, as assessed by dose interruptions, dose reductions, and dose intensity, and study treatment discontinuation because of adverse events | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (63):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Community Cancer Institute (CCI), Fresno, California
  - Baptist - MD Anderson Cancer Center, Jacksonville, Florida
  - University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University Medical Center, Durham, North Carolina
- Australia (6):
  - Prince of Wales Hospital, Randwick, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Monash Health Monash Medical Centre, Clayton, Victoria
  - St Vincent's Hospital Melbourne, Fitzroy, Victoria
  - Peter Maccallum Cancer Centre, Melbourne, Victoria
  - Sir Charles Gairdner Hospital, Nedlands, Western Australia
- Belgium (2):
  - UZ Leuven Gasthuisberg, Leuven
  - CHU de Liège (Sart Tilman), Liège
- China (8):
  - Peking University Third Hospital, Beijing
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Fudan University Shanghai Cancer Center, Shanghai
  - Tianjin Cancer Hospital, Tianjin
  - Wuhan Union Hospital Tongji Medical College, Huazhong University of Science and Technology, Wuhan
  - Zhejiang Cancer Hospital, Zhejiang
  - Henan Cancer Hospital, Zhengzhou
- Denmark (2):
  - Aarhus Universitetshospital Skejby, Aarhus N
  - Rigshospitalet, København Ø
- France (6):
  - Institut Bergonie, Bordeaux
  - Hopital Henri Mondor, Créteil
  - Hopital Claude Huriez, Lille
  - Chu de Montpellier-St Eloi, Montpellier
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - CHU Pontchaillou, Rennes
- Germany (3):
  - Universitatsklinikum Frankfurt, Frankfurt
  - Universitätsklinikum Gießen und Marburg GmbH Standort Gießen Medizinische Klinik I, Giessen
  - Universitaetsklinikum Regensburg, Regensburg
- Poland (5):
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Onkologii Ziemi Lubelskiej im. ?w. Jana z Dukli, Lublin
  - Oddzial Kliniczny Hematologii SPZOZ MSWiA z Warminsko-Mazurskim Centrum Onkologii w Olsztynie, Olsztyn
  - Instytut Hematologii i Transfuzjologii, Warsaw
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroc?aw
- South Korea (6):
  - Pusan National University Hospital, Busan
  - National Cancer Center, Goyang-si
  - Seoul National University Bundang Hospital, Seongnam-si
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic i Provincial, Barcelona
  - Hospital Universitario la Paz, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clinico Universitario de Valencia, Valencia
- Switzerland (2):
  - Inselspital Bern, Insel-Gruppe AG, Bern
  - Universitätsspital Zürich, Zurich
- Taiwan (3):
  - Chang Gung Medical Foundation - Kaohsiung;Oncology, Kaoisung
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
  - Taichung Veterans General Hospital, Xitun Dist.
- United Kingdom (5):
  - Beatson West of Scotland Cancer Centre, Glasgow
  - St James's Institute of Oncology, Leeds
  - UCLH - Clinical Trials Pharmacy B&D Centre, London
  - Christie Hospital, Manchester
  - Nottingham City Hospital, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing

REFERENCES:
- [Derived] Sam J, Leclercq-Cohen G, Gebhardt S, Surowka M, Herter S, Lechner K, Relf J, Briner S, Varol A, Appelt B, Domocos I, Nicolini V, Bez M, Bommer E, Jenni S, Schoenle A, Le Clech M, Colombetti S, Klein C, Umana P, Lundberg P, Korfi K, Bottos A, Bacac M. Preclinical advances in glofitamab combinations: a new frontier for non-Hodgkin lymphoma. Blood. 2025 Oct 9;146(15):1824-1836. doi: 10.1182/blood.2025028863. PMID 40749164
- [Derived] Abramson JS, Ku M, Hertzberg M, Huang HQ, Fox CP, Zhang H, Yoon DH, Kim WS, Abdulhaq H, Townsend W, Herbaux C, Zaucha JM, Zhang QY, Chang H, Liu Y, Cheah CY, Ghesquieres H, Simko S, Orellana-Noia V, Ta R, Relf J, Dixon M, Kallemeijn M, Mulvihill E, Huang H, Lundberg L, Gregory GP. Glofitamab plus gemcitabine and oxaliplatin (GemOx) versus rituximab-GemOx for relapsed or refractory diffuse large B-cell lymphoma (STARGLO): a global phase 3, randomised, open-label trial. Lancet. 2024 Nov 16;404(10466):1940-1954. doi: 10.1016/S0140-6736(24)01774-4. PMID 39550172